CLINICAL TRIAL: NCT02552758
Title: The Influence of Omega-3 Fatty Acid on the Violence of Schizophrenia Patient and the Possible Mechanism
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Mental Health Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2014-25
Record Dates: First submitted 2015-09-08; First posted 2015-09-17 (Estimated); Last update posted 2015-09-17 (Estimated); Status verified 2015-09

CONDITIONS: Schizophrenia
Keywords: violence; PET; omega-3 fatty acid; schizophrenia; patient
MeSH Terms: conditions — Schizophrenia | interventions — Fatty Acids, Omega-3; Positron-Emission Tomography

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Omega-3 fatty acid (Experimental): omega-3 fatty acid
  Interventions: Biological: omega-3 fatty acid; Device: positron emission tomography (PET)
- placebo (Placebo Comparator): placebo
  Interventions: Biological: placebo; Device: positron emission tomography (PET)

INTERVENTIONS:
Biological: omega-3 fatty acid — omega-3 fatty acid
  Arms: Omega-3 fatty acid
Biological: placebo — placebo
  Arms: placebo
Device: positron emission tomography (PET)

SUMMARY:
Investigators plan to explore whether Omega-3 fatty acid have effect on the violent behavior of the schizophrenia patients. Investigators will use PET to explore the influence on serotonin function of the brain to understand the mechanism of how Omega-3 fatty acid works. This study will enroll 100 patients of schizophrenia with violent behavior.Participants will be split into two groups randomly. In one group, participants will receive one pill of placebo per day, and in the other, participants will have one pill of 900mg Omega-3 fatty acid per day. This intervention will last 3 months.At week 0, week 4, week 8 and week 12, some scales will be evaluated. Meanwhile, the density of eicosapentaenoic acid(EPA),docosahexaenoic acid (DHA),noradrenalin(NE), dopamine(DA) and serotonin(5-HT) in blood will be tested.At week 0 and week 12, 10 patients of each group will be randomly selected to have the exam of PET.

ELIGIBILITY:
Inclusion Criteria:

* the sore of MOAS scale >=4 more than 2 violent behavior in recent 6 months by self repot

Exclusion Criteria:

* serious diseases,such as cardiovascular diseases,nervous system disease. allergy to fish oil

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
violent behavior of Participants as Assessed by Modified Overt Aggression Scale(MOAS) | up to 24 months
  change in violent behavior of participants
psychiatry symptoms of participants as assessed by Positive and Negative Syndrome Scale (PANSS) | up to 24 months
  change in psychiatry symptoms of participants
blood level of eicosapentaenoic acid(EPA), docosahexaenoic acid (DHA), noradrenalin(NE), dopamine(DA) and serotonin(5-HT) of participants | up to 24 months
  change in the blood level of DHA, EPA, 5-HT, DA and NE at baseline, 4 weeks, 8 weeks and 12 weeks
the density of 5-HT1A receptor in brain tested by positron emission tomography (PET) | up to 24 months
  change of the density of 5-HT1A receptor in different groups

CONTACTS AND LOCATIONS:
Overall Officials: Yi Qiao, phD, Principal Investigator — Shanghai Mental Health Center (China)
Locations (1):
- Shanghai Mental Health Center, Shanghai, Shanghai Municipality, China